CLINICAL TRIAL: NCT02228122
Title: The Effect of Aquacel® Ag+ Extra Dressing on Wound Biofilms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr Angela Oates (Other)
Collaborators: ConvaTec Inc. (Industry)
Responsible Party: Sponsor-Investigator, Dr Angela Oates, Dr, University of Manchester
Organization: University of Manchester (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UoM Study REF: 14118
Record Dates: First submitted 2014-08-26; First posted 2014-08-28 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-12

CONDITIONS: Diabetes; Chronic Foot Wounds
Keywords: Chronic wounds; Biofilms; Bacteria
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Aquacel® Ag+ Extra (Experimental)
  Interventions: Device: Aquacel® Ag+ Extra

INTERVENTIONS:
Device: Aquacel® Ag+ Extra — Aquacel® Ag+ Extra dressing will be applied to wounds as per instructions for use, dressing to be changed at least one per week for 4 weeks.

SUMMARY:
The purpose of the research is to assess the effects of Aquacel Ag+ Extra dressing on chronic wound bacterial biofilms

DETAILED DESCRIPTION:
Background: Chronic wounds and wound infections can be costly, resulting in prolonged hospital stays and an increased risk of secondary infection and septicaemia. In the UK the management of chronic venous leg ulcers is estimated to cost £1 billion/year, with surgical site infections requiring approximately 6.5 days additional hospital stay. Chronic wounds typically harbour a wide variety of bacteria; heavy bacterial colonisation and subsequent biofilm formation has been cited as a factor which induces a chronic inflammatory state and delays healing times.

AQUACEL®Ag+ Extra is a soft conformable flat sheet nonwoven fabric dressing, which forms a gel when it becomes wet. Its physical characteristics have the potential to increase the speed of antimicrobial action of silver and its effectiveness against any recalcitrant wound bioburden. Removing these potential barriers to healing may help towards wound progression.

Aim: This is a pilot study to investigate the effects of Aquacel Ag+ Extra dressing on chronic wound bacterial biofilms. Wound debridement tissue will be assessed for the presence/absence of in situ biofilms which will be monitored over 4 weeks and compared to the baseline (non-treatment) sample. Additionally, we will evaluate reductions in wound volume over the treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Provided written informed consent
* Be over 18 years of age
* Must have a chronic foot wound greater than 4 weeks in duration
* Be willing and able to attend the clinic for the required study visits -

Exclusion Criteria:

* Subjects with a history of sensitivity to any one of the components of the device being studied
* Subjects who have any other medical condition which, according to the investigator justifies exclusion from the study
* Subjects who are currently participating in or have been on a clinical study within the last 4 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
A measure of the presence/absence of biofilms in over five weeks when exposed to Aquacel Ag+ Extra dressing. | up to day 28
  Wound debridement tissue derived from standard of care will be retained for analysis up to Day 28. Tissue to be sectioned and analysed for the presence or absence of bacterial biofilms.

SECONDARY OUTCOMES:
Size of the wound and an indicator of healing | up to day 28
  Weekly measurements of wound size

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J McBain, BSc, PhD, Principal Investigator — University of Manchester; Angela Oates, BSc, MSc, PhD, FIBMS, Principal Investigator — University of Manchester
Locations (1):
- Manchester Diabetes Centre, Manchester, United Kingdom